CLINICAL TRIAL: NCT03455647
Title: Enhancing Milk Quality and Consumption for Improved Income and Nutrition in Rwanda
Brief Title: Enhancing Milk Consumption for Improved Nutrition in Rwanda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: The International Livestock Research Institute (ILRI) (Other); University of Rwanda (Other); TechnoServe (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0215801
Record Dates: First submitted 2018-02-28; First posted 2018-03-06 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2020-03

CONDITIONS: Inadequate Child Growth
Keywords: stunting; underweight; wasting
MeSH Terms: conditions — Growth Disorders; Thinness; Cachexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ASF Promotion plus Girinka (Experimental): Participants have received a cow from the government of Rwanda through the Girinka program and will receive an animal source food promotion intervention from the study.
  Interventions: Behavioral: ASF promotion plus Girinka
- Girinka only (No Intervention): Participants have received a cow from the government of Rwanda through the Girinka program and will not receive any intervention from the study.
- Girinka eligible (No Intervention): Participants are eligible to receive a cow through the government of Rwanda Girinka program, but have not yet received a cow. They will not receive any intervention from the study.

INTERVENTIONS:
Behavioral: ASF promotion plus Girinka — Behavior change communication promoting the consumption of milk produced in the household and other optimal maternal and child nutrition practices. The intervention will be implemented by government of Rwanda Community Health Workers.
  Arms: ASF Promotion plus Girinka

SUMMARY:
This study is a mixed-methods cluster-randomized controlled trial in Rwanda designed to measure the impact of a dairy asset transfer program with or without nutrition education promoting the home consumption of dairy milk and other animal source foods.

DETAILED DESCRIPTION:
The purpose of this research is to contribute to efforts for improving the consumption of milk in Rwanda. It will do so by generating and communicating evidence on the nutritional benefits of including animal source food (ASF) in diets of young children and pregnant and lactating women through nutrition education. The proposed project draws upon the work of a Government of Rwanda program - the One Cow per Poor Family (Girinka) program. The Girinka program (2006 - present) is a country-wide program whose goal is to increase household income and reduce child malnutrition among poor households through livestock asset transfer. The study has two main objectives. First, researchers will measure the impact of a nutrition education/ASF promotion intervention on child and maternal nutritional status in households that have received a cow through the Girinka program. Second, researchers will compare nutrition outcomes in the Girinka + nutrition education and Girinka only groups to individuals in households that are eligible for Girinka, but have not yet received a cow. The nutrition education/ASF promotion intervention will be designed and overseen by a local organization and implemented through Government of Rwanda community health workers. The main study outcomes are child height-for-age z-score, child milk consumption, and child dietary diversity. The secondary outcomes are child weight-for-age z-score, child weight-for-height z-score, and maternal body-mass index. The researchers plan to randomly assign all cells in two districts to receive the nutrition education intervention or no intervention. The study will enroll a cohort of 687 mother-child pairs (229 per study arm). The aim is to enroll children 12-17 months of age at baseline; however, if there are not adequate numbers of households that meet all other eligibility criteria, then the child age range will be expanded to 12-29 months of age at baseline. The research team will conduct baseline and endline surveys to measure differences between the groups. At endline, researchers will collect qualitative data from participants and community health workers in the intervention arm to triangulate with the survey findings.

ELIGIBILITY:
Inclusion Criteria:

Arm 1:

* Household is located in an intervention cell
* Household received a cow under the government of Rwanda Girinka program before 2017
* Household contains a mother 18-49 years of age
* Household contains a child between the ages of 12 and 29 months at baseline

Arm 2:

* Household is located in a comparison cell
* Household received a cow under the government of Rwanda Girinka program before 2017
* Household contains a mother 18-49 years of age
* Household contains a child between the ages of 12 and 29 months at baseline

Arm 3:

-- Household is located in a comparison cell

* Household is eligible to receive a cow under the government of Rwanda Girinka program
* Household contains a mother 18-49 years of age
* Household contains a child between the ages of 12 and 29 months at baseline

Exclusion Criteria:

* Failure to meet inclusion criteria

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The target population is mothers with a child between the ages of 12 and 29 months at study initiation. The child may be male or female.
Enrollment: 746 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Child height-for-age z-score (HAZ) | Baseline at study initiation
  Measure child recumbent length in triplicate and age reported by mother. HAZ will be calculated using the World Health Organization standard.
Child height-for-age z-score (HAZ) | Endline (approximately one year)
  Measure child recumbent length in triplicate and age reported by mother. HAZ will be calculated using the World Health Organization standard.
Child dairy milk consumption | Baseline at study initiation
  Measurement based on 24 hour recall of consumption amount
Child milk consumption | Endline (approximately one year)
  Measurement based on 24 hour recall of consumption amount
Child dietary diversity | Baseline at study initiation
  Measurement based on 24 hour recall of consumption and calculated using the World Health Organization child dietary diversity indicator
Child dietary diversity | Endline (approximately one year)
  Measurement based on 24 hour recall of consumption and calculated using the World Health Organization child dietary diversity indicator

SECONDARY OUTCOMES:
Child weight-for-height z-score (WHZ) | Baseline at study initiation
  Measurement based on recumbent length and body weight measured in triplicate. WHZ will be calculated using the World Health Organization standard.
Child weight-for-height z-score (WHZ) | Endline (approximately one year)
  Measurement based on recumbent length and body weight measured in triplicate. WHZ will be calculated using the World Health Organization standard.
Child weight for age z-score (WAZ) | Baseline at study initiation
  Measurement based on weight measured in triplicate and age reported by mother. WAZ will be calculated based on the World Health Organization standard.
Child weight for age z-score (WAZ) | Endline (approximately one year)
  Measurement based on weight measured in triplicate and age reported by mother. WAZ will be calculated based on the World Health Organization standard.
Maternal body-mass index | Baseline at study initiation
  Measurement based on weight and standing height.
Maternal body-mass index | Endline (approximately one year)
  Measurement based on weight and standing height.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Flax, PhD, MPH, Principal Investigator — RTI International
Locations (2):
- Rwanda (2):
  - Ruhango District, Ruhango, Southern Province
  - Nyabihu District, Nyabihu, Western Province

IPD SHARING:
Plan to Share IPD: Yes